CLINICAL TRIAL: NCT05147233
Title: A Randomized, Double-masked, Vehicle-controlled Study Evaluating the Efficacy and Safety of OCS-01 Eyedrops Compared to Vehicle in the Treatment of Inflammation and Pain Following Cataract Surgery
Brief Title: A Phase 3 Study Evaluating the Efficacy and Safety of OCS-01 Eyedrops Compared to Vehicle for the Treatment of Ocular Inflammation and Pain Following Cataract Surgery
Acronym: OPTIMIZE-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Oculis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DX218
Record Dates: First submitted 2021-11-24; First posted 2021-12-07 (Actual); Results first posted 2025-07-11 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-05

CONDITIONS: Inflammation Eye Pain; Postoperative Cataract

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- OCS-01 (Experimental): 1 drop of OCS-01 (Dexamethasone ophthalmic suspension 1.5% [15 mg/mL]) in the study eye once daily (QD) for 14 days, beginning 1-day post-surgery in the study eye.
  Interventions: Drug: OCS-01
- Vehicle (Placebo Comparator): 1 drop of vehicle in the study eye QD for 14 days, beginning 1-day post-surgery in the study eye.
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: OCS-01 — Dexamethasone ophthalmic suspension, 1.5%
  Arms: OCS-01
Drug: Vehicle — Vehicle
  Arms: Vehicle

SUMMARY:
This was a randomized, double-masked, vehicle-controlled, Phase 3 study evaluating the efficacy and safety of OCS-01 QD compared to vehicle in the treatment of inflammation and pain following cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

* Be planning to undergo unilateral cataract extraction via phacoemulsification and posterior chamber intraocular lens (PCIOL) implantation in the study eye.
* Have a pin-hole visual acuity (VA) without any other correction > 20 letters (approximately 20/400) in the operative eye and > 35 letters (approximately 20/200) in the fellow eye as measured using an Early Treatment for Diabetic Retinopathy Study (ETDRS) chart at Visit 1 (Day -1 to Day -28 [prior to surgery]).

Exclusion Criteria:

* Have any intraocular inflammation (e.g. white blood cells or flare) present in either eye at the Visit 1 (Day -1 to Day -28 [prior to surgery]) slit lamp examination.
* Have a score > 0 on the Ocular Pain Assessment at Visit 1 (Day -1 to Day -28 [prior to surgery]) in the study eye.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 241 (Actual)
Dates: Start 2022-06-24 (Actual); Primary Completion 2023-06-22 (Actual); Study Completion 2023-07-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (25):
- United States (25):
  - Oculis Site 16, Chandler, Arizona
  - Oculis Site 28, Phoenix, Arizona
  - Oculis Site 8, Fayetteville, Arkansas
  - Oculis Site 9, Inglewood, California
  - Oculis Site 23, Newport Beach, California
  - Oculis Site 26, Petaluma, California
  - Oculis Site 24, San Pedro, California
  - Oculis Site 22, Westminster, California
  - Oculis Site 11, Fort Collins, Colorado
  - Oculis Site 12, Tamarac, Florida
  - Oculis Site 17, Morrow, Georgia
  - Oculis Site 20, Louisville, Kentucky
  - Oculis Site 5, St Louis, Missouri
  - Oculis Site 3, Washington, Missouri
  - Oculis Site 13, Kinston, North Carolina
  - Oculis Site 6, Brecksville, Ohio
  - Oculis Site 14, Cincinnati, Ohio
  - Oculis Site 25, Eugene, Oregon
  - Oculis Site 7, Kingston, Pennsylvania
  - Oculis Site 4, Austin, Texas
  - Oculis Site 10, Houston, Texas
  - Oculis Site 2, San Antonio, Texas
  - Oculis Site 31, San Antonio, Texas
  - Oculis Site 27, Salt Lake City, Utah
  - Oculis Site 30, Lynchburg, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- OCS-01: 1 drop of OCS-01 in the study eye once QD for 14 days, beginning 1-day post-surgery in the study eye.
- Vehicle: 1 drop of vehicle in the study eye once QD for 14 days, beginning 1-day post-surgery in the study eye.
Period: Overall Study
Arm/Group | OCS-01 | Vehicle
Started | 119 | 122
Completed | 116 | 118
Not Completed | 3 | 4
Not completed — Adverse Event | 0 | 1
Not completed — Lost to Follow-up | 1 | 1
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 2 | 1

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) consists of all randomized subjects who were analyzed under the treatment to which they were randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | OCS-01 | Vehicle | Total
Number analyzed (Participants) | 119 | 122 | 241
Age, Continuous [Mean (Standard Deviation); unit: Years] | 68.8 (7.80) | 67.8 (8.98) | 68.3 (8.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71 | 70 | 141
  Male | 48 | 52 | 100
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 26 | 26 | 52
  Not Hispanic or Latino | 93 | 96 | 189
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 6 | 5 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 17 | 25 | 42
  White | 95 | 91 | 186
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Absence of Anterior Chamber Cells at Visit 6.
Time Frame: Day 15
Population: FAS
Measure: Number; unit: percentage of study eyes
Units Other Than Participants: study eye
Groups:
- OCS-01; Vehicle: 1 drop of OCS-01 in the study eye QD for 14 days, beginning 1-day post-surgery in the study eye.
Arm/Group | OCS-01 | Vehicle
Number analyzed (Participants) | 119 | 122
Number analyzed (study eye) | 119 | 122
percentage of study eyes | 57.2 | 24.0
Statistical Analysis 1: Comparison: OCS-01 vs Vehicle; Test type: Superiority; p < 0.0001, Wald test; Difference in Percentages = 33.2, 95% CI 2-sided [21.5 to 44.9]

2. Primary Outcome: Absence of Ocular Pain at Visit 4.
Time Frame: Day 4
Population: FAS
Measure: Number; unit: percentage of study eyes
Units Other Than Participants: study eye
Arm/Group | OCS-01 | Vehicle
Number analyzed (Participants) | 119 | 122
Number analyzed (study eye) | 119 | 122
percentage of study eyes | 75.5 | 52.0
Statistical Analysis 1: Comparison: OCS-01 vs Vehicle; Test type: Superiority; p < 0.0001, Wald test; Difference in Percentages = 23.5, 95% CI 2-sided [11.7 to 35.3]

ADVERSE EVENTS:
Time Frame: From first dose until Day 90
Arm/Group | OCS-01 | Vehicle
All-Cause Mortality (participants affected / at risk) | 0/119 | 0/122
Serious Adverse Events (participants affected / at risk) | 0/119 | 1/122
Other Adverse Events (participants affected / at risk) | 2/119 | 8/122
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OCS-01 (N=119) | Vehicle (N=122)
Covid-19 (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OCS-01 (N=119) | Vehicle (N=122)
Eye Pain (Eye disorders) | 2 (2) | 8 (8) — Study eye

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2022-05-10): https://cdn.clinicaltrials.gov/large-docs/33/NCT05147233/Prot_000.pdf
  • Statistical Analysis Plan (2023-07-13): https://cdn.clinicaltrials.gov/large-docs/33/NCT05147233/SAP_001.pdf